CLINICAL TRIAL: NCT06007781
Title: A Phase 1, Randomized, Double-blind, Multi-center, Placebo-controlled Trial to Evaluate the Safety and Immunogenicity of the Intramuscular Norovirus GI.1/GII.4 Bivalent VLP Vaccine in Healthy Japanese Infants 5 Months of Age at First Trial Vaccine Administration
Brief Title: Safety and Immunogenicity of HIL-214 in Healthy Japanese Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HilleVax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-109
Record Dates: First submitted 2023-08-15; First posted 2023-08-23 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Intervention Model Description: Subjects will be allocated (2 to1) into one of two trial arms, Arm 1 - One dose of HIL-214; Arm 2 - One dose of placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): One dose of placebo on Day 1 and one dose of placebo between Day 29 and Day 57
  Interventions: Biological: Placebo
- Experimental (Experimental): One dose of HIL-214 on Day 1 and one dose of HIL-214 between Day 29 and Day 57
  Interventions: Biological: HIL-214

INTERVENTIONS:
Biological: Placebo — 2 injections - given on Day 1 and the second given between Day 29 - Day 57
  Arms: Placebo
Biological: HIL-214 — 2 injections - given on Day 1 and the second given between Day 29 - Day 57
  Arms: Experimental

SUMMARY:
This is a phase 1, randomized, double-blind multi-center, placebo-controlled trial in Japan to evaluate the safety and immunogenicity of HIL-214 in healthy infants 5 months of age (-14/+14 days) at first trial vaccine administration. In this protocol, because the trial is blinded, trial vaccine refers to both the investigational vaccine (HIL-214) and placebo.

DETAILED DESCRIPTION:
The rationale for trial NOR-109 is to evaluate the safety and immunogenicity of HIL-214 in Japanese pediatric subjects and establish whether the data obtained is consistent with that previously obtained for non-Japanese pediatric subjects.

The clinical trials for HIL-214 have so far been performed in Europe, the United States and several countries in Latin America [26]. The incidence rate of norovirus-attributable disease in Japan is at least as high as in other developed countries with the highest rates occurring in children below the age of 5 years and hospitalization most common in very young and very old populations. The inclusion of infants (5 months [±14 days] of age at the time of first trial vaccine administration) serves to compare the data obtained for infants of non-Japanese descent with Japanese infants, in alignment with the global clinical program, and to support the inclusion of Japanese infants into phase 3. Enrollment and vaccination of the infants will be performed either before or after the required routine childhood vaccines per the national immunization schedule.

This phase 1 trial in Japan aims to assess the safety and immunogenicity of two doses of HIL-214 administered 4 to 8 weeks apart, in 21 healthy infants aged 5 months at the time of the first trial vaccine dose administration. A placebo arm is included to allow an unbiased assessment of safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria

* Male or female subject aged 5 months [-14/+14 days].
* Infants who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
* The subject's legally acceptable representative (LAR) signs and dates a written, informed consent form (ICF) and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
* The subject's LAR is willing and able to comply with trial procedures and is available for the duration of follow-up.

Exclusion Criteria

* Clinically significant abnormality in growth by length/height, weight, or head circumference (according to national guidelines).
* Gastrointestinal abnormalities or any chronic gastrointestinal disease, including any uncorrected congenital malformation of the gastrointestinal tract according to medical history and/or physical examination.
* Chronic use of oral corticosteroids (equivalent to 20 mg/day prednisolone for ≥12 weeks / ≥2 mg/kg body weight /day for ≥2 weeks) within 60 days prior to Visit 1 (use of inhaled, intranasal, or topical corticosteroids are allowed).
* Use of parenteral corticosteroids (equivalent to 20 mg/day prednisolone for ≥12 weeks / ≥2 mg/kg body weight /day for ≥2 weeks. Use of inhaled, intranasal, or topical corticosteroid is allowed) within 60 days prior to Visit 1.
* Receipt of immunostimulants within 60 days prior to Visit 1.
* Receipt of parenteral, epidural, or intra-articular immunoglobulin (Ig) preparations, blood products, and/or plasma derivatives within 90 days prior to Visit 1 or planned during the full duration of the trial.
* Receipt of immunosuppressive therapy prior to Visit 1.
* Known hypersensitivity or allergy to any of the trial vaccine components (including excipients).
* Any clinically significant active infection (as assessed by the investigator) or temperature ≥38.0°C (>100.4°F), regardless of method used, within 3 days prior to intended trial vaccine administration.
* Gastroenteritis within 7 days before planned dosing (can warrant delay of trial vaccine administration).
* History of, e.g., convulsions/febrile convulsions, or any illness, that, in the opinion of the investigator, might interfere with the results of the trial or pose additional risk to the subjects due to participation the trial.
* Abnormalities of splenic or thymic function.
* Known or suspected impairment/alteration of immune function.
* Known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Receipt or scheduled receipt of any other approved or authorized vaccines within 14 days (for all non-live vaccines or oral live vaccines) or 28 days (for parenteral live vaccines) before or after trial vaccine administration.
* Participation in any clinical trial with another investigational product 30 days prior to first trial visit or intention to participate in another clinical trial at any time during the conduct of this trial.
* Seropositive for, or in evaluation for, possible human immunodeficiency virus infection.

Ages: 5 Months to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Fukui Aiiku Hospital, Fukui-shi
  - Iizuka Children's Clinic, Iizuka-Shi
  - Childrens Clinic of Kose, Kofu
  - Ohigesenseino Kodomo Clinic, Sapporo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the trial at 4 investigative sites in Japan from 18 August 2023 to 27 May 2024
Pre-assignment Details: Participants were enrolled in 1 of 2 treatment arms and received 2 doses of either HIL-214, a norovirus vaccine comprising 50 µg GI.1 virus-like particle (VLP) and 150 µg GII.4c VLP, adjuvanted with 500 µg of aluminum hydroxide, or placebo.
Groups:
- HIL-214: One dose of HIL-214 on Day 1 and one dose of HIL-214 between Day 29 and Day 57
Period: Overall Study
Arm/Group | Placebo | HIL-214
Started | 7 | 14
Completed | 7 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, all participants that received trial vaccine (HIL-214 or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | HIL-214 | Total
Number analyzed (Participants) | 7 | 14 | 21
Age, Continuous [Mean (Standard Deviation); unit: days] | 152.9 (7.60) | 150.9 (7.72) | 151.6 (7.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 14 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 14 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 7 | 14 | 21
Weight [Mean (Standard Deviation); unit: kg] | 7.23 (0.596) | 7.31 (0.815) | 7.29 (0.735)
Length [Mean (Standard Deviation); unit: cm] | 63.96 (1.936) | 64.27 (2.083) | 64.17 (1.992)
Head circumference [Mean (Standard Deviation); unit: cm] | 41.86 (1.282) | 41.66 (1.873) | 41.73 (1.668)

OUTCOME MEASURES:

1. Primary Outcome: Safety of HIL-214 Compared to Placebo - AEs Leading to Trial Withdrawal
Description: Percentage of Participants with Adverse Events (AEs) Leading to Trial Withdrawal
Time Frame: Day 1 to 6 months post-dose 2
Population: Safety Analysis Set, all participants that received trial vaccine (HIL 214 or placebo).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 7 | 14
Percentage of Participants | 0 | 0

2. Primary Outcome: Safety of HIL-214 Compared to Placebo - Solicited Local Adverse Events
Description: Percentage of Participants with Solicited Local (Injection Site) Adverse Events (AEs) Within 7 Days of Vaccine Administration (any dose). Assessed AEs included pain, erythema, induration, and swelling.
Time Frame: Day 1 to Day 7 post-dose 1 and Day 1 to Day 7 post-dose 2 (Day 36 to Day 56)
Population: Safety Analysis Set, all participants that received trial vaccine (HIL 214 or placebo).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 7 | 14
Percentage of Participants
  Any solicited local AE | 0 | 42.9
  Pain | 0 | 14.3
  Erythema | 0 | 14.3
  Induration | 0 | 14.3
  Swelling | 0 | 14.3

3. Primary Outcome: Safety of HIL-214 Compared to Placebo - Solicited Systemic Adverse Events
Description: Percentage of Participants with Solicited Systemic Adverse Events (AEs) Within 7 Days of Vaccine Administration. Assessed AEs included drowsiness, irritability/fussiness, loss of appetite, fever, vomiting, and diarrhea.
Time Frame: Day 1 to Day 7 post-dose 1 and Day 1 to Day 7 post-dose 2 (Day 36 to Day 56)
Population: Safety Analysis Set, all participants that received trial vaccine (HIL 214 or placebo).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 7 | 14
Percentage of Participants
  Any solicited systemic AE | 14.3 | 64.3
  Drowsiness | 14.3 | 35.7
  Irritability/fussiness | 0 | 35.7
  Loss of appetite | 0 | 21.4
  Fever | 0 | 7.1
  Vomiting | 0 | 21.4
  Diarrhea | 0 | 35.7

4. Primary Outcome: Safety of HIL-214 Compared to Placebo - Percentage of Participants With AEs Leading to Vaccine Withdrawal
Description: Percentage of participants with AEs that lead to withdrawal of trial vaccine up to the planned time of second dose administration.
Time Frame: Up to 56 days post-dose 1
Population: Safety Analysis Set, all participants that received trial vaccine (HIL 214 or placebo).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 7 | 14
Percentage of Participants | 0 | 0

5. Secondary Outcome: Immunogenicity of HIL-214 Compared to Placebo.
Description: The percentage of participants with a predefined seroresponse (≥4-fold rise in antibody concentration) at Visit 2, Visit 3, and/or Visit 4 to the GI.1 and GII.4c components of HIL-214 and 95% confidence interval are reported. HBGA-blocking and pan-Ig assays were used for immunogenicity analyses.
Time Frame: Day 1 to 6 months post-dose 2
Population: Per-Protocol Set, all participants who received trial vaccine (HIL-214 or placebo) and had no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | HIL-214
Number analyzed (Participants) | 7 | 13
Percentage of Participants
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 2: number analyzed (Participants) | 7 | 8
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 2 | 0 [0.0 to 41.1] | 87.5 [47.3 to 99.7]
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 3: number analyzed (Participants) | 7 | 12
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 3 | 0 [0.0 to 41.1] | 100 [73.5 to 100.0]
  Anti-GI.1 HBGA-blocking seroresponse rate at Visit 4 | 0 [0.0 to 41.1] | 100 [73.5 to 100.0]
  Anti-GII.4c HBGA-blocking seroresponse rate at Visit 2 | 0 [0.0 to 41.1] | 23.1 [5.0 to 53.8]
  Anti- GII.4c HBGA-blocking seroresponse rate at Visit 3 | 0 [0.0 to 41.1] | 92.3 [64.0 to 99.8]
  Anti- GII.4c HBGA-blocking seroresponse rate at Visit 4 | 28.6 [3.7 to 71.0] | 84.6 [54.6 to 98.1]
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 2: number analyzed (Participants) | 7 | 8
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 2 | 0 [0.0 to 41.1] | 37.5 [8.5 to 75.5]
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 3: number analyzed (Participants) | 7 | 12
  Anti-GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 3 | 0 [0.0 to 41.1] | 91.7 [61.5 to 99.8]
  Anti- GI.1 and GII.4c HBGA-blocking seroresponse rate at Visit 4 | 0 [0.0 to 41.1] | 84.6 [54.6 to 98.1]
  Anti-GI.1 pan-Ig seroresponse rate at Visit 2 | 0 [0.0 to 41.1] | 100 [75.3 to 100.0]
  Anti-GI.1 pan-Ig seroresponse rate at Visit 3 | 0 [0.0 to 41.1] | 100 [75.3 to 100.0]
  Anti-GI.1 pan-Ig seroresponse rate at Visit 4 | 0 [0.0 to 41.1] | 100 [75.3 to 100.0]
  Anti-GII.4c pan-Ig seroresponse rate at Visit 2 | 0 [0.0 to 41.1] | 69.2 [38.6 to 90.9]
  Anti-GII.4c pan-Ig seroresponse rate at Visit 3 | 0 [0.0 to 41.1] | 100 [75.3 to 100.0]
  Anti-GII.4c pan-Ig seroresponse rate at Visit 4 | 28.6 [3.7 to 71.0] | 84.6 [54.6 to 98.1]
  Anti-GI.1 and GII.4c pan-Ig seroresponse rate at Visit 2 | 0 [0.0 to 41.1] | 69.2 [38.6 to 90.9]
  Anti-GI.1 and GII.4c pan-Ig seroresponse rate at Visit 3 | 0 [0.0 to 41.1] | 100 [75.3 to 100.0]
  Anti- GI.1 and GII.4c pan-Ig seroresponse rate at Visit 4 | 0 [0.0 to 41.1] | 84.6 [54.6 to 98.1]

ADVERSE EVENTS:
Time Frame: Serious adverse events from Day 1 to 6 months post-dose 2; Unsolicited adverse events from Day 1 to 28 days post-dose 1 and Day 1 to 28 days post-dose 2.
Arm/Group | Placebo | HIL-214
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/14
Other Adverse Events (participants affected / at risk) | 7/7 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | HIL-214 (N=14)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Bloody stool
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) — Worsening of gastroenteritis norovirus
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | HIL-214 (N=14)
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT06007781/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT06007781/SAP_001.pdf